CLINICAL TRIAL: NCT05277831
Title: Testing the Efficacy of A Scalable, Telephone-Delivered, Guided Imagery Tobacco Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Judith S. Gordon, PhD, Professor and Associate Dean for Research, University of Arizona
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2103633455; R01AT011500 (NIH)
Record Dates: First submitted 2022-02-14; First posted 2022-03-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Smoking; Smoking Reduction; Smoking, Cigarette; Smoking (Tobacco) Addiction; Smoking Habit
MeSH Terms: conditions — Smoking Cessation; Smoking; Smoking Reduction; Cigarette Smoking; Behavior, Addictive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery Intervention (Experimental): Guided Imagery Intervention
  Interventions: Other: Guided Imagery Intervention
- Standard Behavioral Control (Active Comparator): Standard Behavioral Control
  Interventions: Other: Standard Behavioral Control

INTERVENTIONS:
Other: Guided Imagery Intervention — Participants in the Guided Imagery Intervention receive 6 sessions of a Guided Imagery plus standard smoking cessation coaching over 6 weeks, delivered by telephone. Sessions range from 10 - 60 minutes, and cover reasons for and benefits of quitting, triggers and alternative strategies, coping with cravings, withdrawal and NRT, and relapse prevention. In each session, coaches work with participants to create or revise guided imagery scripts. After the session, coaches record the script as a digital audio file and send to the participant. Participants listen to their audio file every day and practice behavioral skills between sessions.
  Arms: Guided Imagery Intervention
Other: Standard Behavioral Control — Participants in the Standard Behavioral Control condition receive 6 sessions of a standard smoking cessation coaching over 6 weeks, delivered by telephone. Sessions range from 10 - 60 minutes, and cover reasons for and benefits of quitting, triggers and alternative strategies, coping with cravings, withdrawal and NRT, and relapse prevention. In each session, coaches work with participants to identify lifestyle changes to support tobacco cessation, and set a schedule for practicing new behavioral strategies. Participants complete exercises in a quit booklet every day and practice behavioral skills between sessions.
  Arms: Standard Behavioral Control

SUMMARY:
The objective of this R01 application is to conduct a randomized controlled trial to test the efficacy of the Be Smoke Free, telephone-based, guided imagery (GI) intervention (IC) for smoking cessation compared to active behavioral control (CC). The study will recruit 1,200 diverse smokers from three states, Arizona, New York, and West Virginia to increase generalizability. Participants will be randomly assigned to receive either the IC or CC delivered by telephone by University of Arizona study coaches and will be assessed at 3- and 6-months post-enrollment by study staff. The primary outcome is biochemically verified 7-day point prevalence abstinence at 6 months. This innovative and rigorously designed project conducted by an experienced team has the potential to improve public health through the delivery of an innovative integrative GI intervention via telephone.

DETAILED DESCRIPTION:
The Specific Aims of the proposed study are to:

Aim 1: Test the efficacy of a telephone-delivered, integrative GI tobacco cessation intervention (IC) vs. an active behavioral control (CC) on biochemically verified 7-day point prevalence and self-reported 30-day smoking abstinence at 6 months post-enrollment. Four weeks of nicotine replacement therapy (NRT) will be included in both conditions. The investigators will assess self-reported 7-day and 30-day tobacco use at baseline, and 3- and 6-months post-enrollment. Our primary outcome is biochemically verified 7-day point prevalence abstinence at 6 months using the Smokerlyzer iCO expired CO monitor.

H1: Participants in the IC will have 10% higher quit rates than those in the CC. A 10% increase is clinically meaningful on a population level. A sample size of 1200 will provide 90% power to detect a 10% increase over a control condition quit rate of 30% with 20% missing data.

Aim 2: Conduct dose-response analyses on the effect of IC adherence (measured by self-reported minutes of intervention use per week, number of times GI skills practiced per weeks, number of sessions attended, and coach-rated participant engagement in sessions) on abstinence at 6 months. The investigators will also examine effects of the IC and CC on tobacco use for those participants who do not report abstinence at 6-months.

H2A: IC participants who are more adherent will have higher rates of biochemically verified abstinence.

H2B: IC and CC participants who do not report abstinence will report significant reductions in tobacco use.

Aim 3: Conduct subgroup analyses of moderators (e.g., phone type/plan, recruitment method, location, sex, race/ethnicity, level of dependence) on tobacco cessation outcomes at 6 months, and assess participants using a mixed-methods approach (e.g., surveys, in-depth interviews) for exploring sub-group differences. This innovative and rigorously designed project conducted by an experienced team has the potential to improve public health through the delivery of an innovative integrative GI intervention via telephone. If successful, this intervention model could be expanded to address other forms of tobacco and e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Report daily smoking in the last 30 days
* Age 18 or over
* Speak English
* Have a smart phone with internet access
* Willing to receive coaching over the phone

Exclusion Criteria:

* No phone
* No internet access
* Does not speak English
* More than one person per household
* Psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1209 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieve biochemically verified 7 day smoking abstinence | 6 months
  Smoking abstinence will be biochemically verified with expired carbon monoxide

SECONDARY OUTCOMES:
Number of participants who report 7 day smoking abstinence | Baseline, 3 months, and 6 months
  Participants will self-report tobacco use
Number of participants who report 30 day smoking abstinence | Baseline, 3 months, and 6 months
  Participants will self-report tobacco use
Number of minutes of intervention use per week | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  Number of minutes participants engage in study sessions per week
Number of minutes guided imagery and other integrative skills practiced per day | 3 months, 6 months
  Participants will self-report number of minutes guided imagery and other integrative skills practiced per day for the past 7 days
Number of intervention sessions attended | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Gordon JS, Armin JS, Giacobbi P Jr, Hsu CH, Marano K, Sheffer CE. Testing the Efficacy of a Scalable Telephone-Delivered Guided Imagery Tobacco Cessation Treatment: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2023 Jun 23;12:e48898. doi: 10.2196/48898. PMID 37351932